CLINICAL TRIAL: NCT00264550
Title: A Multicenter, Randomized, Double-blind, Placebo-controlledTrial of Golimumab, a Fully Human Anti-TNFa MonoclonalAntibody, Administered Subcutaneously, in Subjects With ActiveRheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: An Efficacy and Safety Study of Golimumab in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Acronym: GO-FORWARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006343; C0524T06 (Other: Centocor); 2004-003296-36 (EudraCT Number)
Record Dates: First submitted 2005-12-11; First posted 2005-12-13 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Golimumab; Methotrexate; Fully Human anti-TNFa monoclonal antibody; Simpony
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Placebo + Methotrexate (Placebo Comparator): Placebo subcutaneous (SC) injections every 4 weeks from Week 0 to Week 20 (early escape at Week 16); Methotrexate - 15 to 25mg weekly from Week 0 up to 5 yrs; Golimumab - if early escape, 50mg SC injections every 4 weeks from Week 16 up to 5 years; Golimumab - 50 mg SC injections every 4 weeks from Week 24 up to 5 yrs (unless early escape); Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100mg and from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Methotrexate; Drug: Placebo injection
- Group 2: Golimumab 100 mg + Placebo (Experimental): Golimumab 100 mg SC injections every 4 weeks from Week 0 up to 5 yrs; Placebo - 7-10 capsules weekly during blinded period (or Week 16 if early escape); Methotrexate - if early escape, 15 to 25mg weekly from Week 16 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Golimumab 100 mg; Drug: Placebo capsules
- Group 3: Golimumab 50 mg + Methotrexate (Experimental): Golimumab 50 mg SC injections every 4 weeks from Week 0 up to 5 yrs (unless early escape at Week 16); Methotrexate - 15 to 25 mg weekly from Week 0 up to 5 years; Golimumab - if early escape, 100 mg SC injections every 4 weeks from Week 16 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to100mg and from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Golimumab 50 mg; Drug: Methotrexate
- Group 4: Golimumab 100 mg + Methotrexate (Experimental): Golimumab100 mg SC injections every 4 weeks from Week 0 up to 5 yrs; Methotrexate - 15 to 25 mg weekly from Week 0 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Golimumab 100 mg; Drug: Methotrexate

INTERVENTIONS:
Drug: Golimumab 100 mg — Participants will receive subcutaneous (SC) injections of golimumab 100 mg every 4 weeks.
  Arms: Group 2: Golimumab 100 mg + Placebo; Group 4: Golimumab 100 mg + Methotrexate
Drug: Golimumab 50 mg — Participants will receive subcutaneous (SC) injections of golimumab 50 mg every 4 weeks.
  Arms: Group 3: Golimumab 50 mg + Methotrexate
Drug: Methotrexate — Participants will receive methotrexate capsules weekly.
  Arms: Group 1: Placebo + Methotrexate; Group 3: Golimumab 50 mg + Methotrexate; Group 4: Golimumab 100 mg + Methotrexate
Drug: Placebo injection — Participants will receive subcutaneous (SC) injections of placebo every 4 weeks.
  Arms: Group 1: Placebo + Methotrexate
Drug: Placebo capsules — Participants will receive placebo capsules weekly
  Arms: Group 2: Golimumab 100 mg + Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of golimumab, alone or in combination with methotrexate (MTX), as compared to methotrexate alone in rheumatoid arthritis (RA) patients who have active rheumatoid arthritis despite treatment with MTX.

DETAILED DESCRIPTION:
This is a randomized (treatment is assigned by chance), double-blind (neither the physician nor the patient is aware of the received treatment), placebo-controlled study of multiple subcutaneous (SC) administrations of golimumab at 2 doses as monotherapy or in combination with MTX in patients with active RA despite treatment with MTX. The duration of participation in the study for an individual patient will be upto 268 weeks. The patients will be randomly assigned in a 3:3:2:2 ratio to receive golimumab 50 mg or 100 mg or placebo injections under the skin every 4 weeks through week 20 and methotrexate or placebo capsules will be given in addition. At Week 24, all subjects will receive golimumab 50mg or 100mg injections, and golimumab continues for all groups for about 4 and a half more years. At Week 16 any patient in the study who meets criteria for < 20% improvement from baseline in both swollen and tender joint count will enter early escape in a double-blinded fashion. Treatment during the long-term extension will start at Week 52 and continue every 4 weeks thereafter for a total of approximately 5 years from the initial (Week 0) administration of study agent. Patients will return for scheduled follow-up visits generally every 12 weeks for a total length of follow-up of approximately 5 years from the first administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) (according to the revised 1987 criteria of the ACR) for at least 3 months prior to screening
* Must have been treated with and tolerated methotrexate (MTX) at a dose of at least 15 mg/week for at least 3 months prior to screening, and have a MTX dose of >=15 mg/week and <=25 mg/week and stable for at least 4 weeks prior to screening
* Have active RA as defined by persistent disease activity with at least 4 swollen and 4 tender joints, at the time of screening and baseline, and at least 2 of the following 4 criteria: a)C-reactive protein (CRP) >=1.5 mg/dL at screening or erythrocyte sedimentation rate (ESR) by Westergren method of >= 28 mm in the first hour at screening or baseline, b)Morning stiffness of >= 30 minutes at screening and baseline, c)Bone erosion by x-ray and/or magnetic resonance imaging (MRI) prior to first administration of study agent, d)Anti-cyclic citrullinated peptide (anti-CCP) antibody-positive or rheumatoid factor (RF) positive at screening
* If using oral corticosteroids, must be on a stable dose equivalent to <= 10 mg of prednisone/day for at least 2 weeks prior to first administration of study agent
* Are considered eligible according to specified tuberculosis (TB) screening criteria

Exclusion Criteria:

* Have inflammatory diseases other than RA that might confound the evaluation of the benefit of golimumab therapy
* Have had treatment with disease-modifying anti-rheumatic drugs (DMARDs)/systemic immunosuppressives other than MTX, during the 4 weeks prior to the first administration of study agent
* Have had prior treatment with biologic anti-tumor necrosis factor (TNF) drugs (infliximab, etanercept, adalimumab)
* Have had history of, or ongoing, chronic or recurrent infectious disease.
* Have serious infection within 2 months prior to first administration of study agent
* Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2005-12; Primary Completion 2007-09 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (50):
- United States (13):
  - Mobile, Alabama
  - Palo Alto, California
  - Pasadena, California
  - Upland, California
  - Ormond Beach, Florida
  - Palm Harbor, Florida
  - Moline, Illinois
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Duncansville, Pennsylvania
  - Richmond, Virginia
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Rosario
  - S.M. de Tucuman
  - San Miguel de Tucumán
- Australia (3):
  - Clayton
  - Maroochydore
  - Melbourne
- Canada (6):
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Ottawa, Ontario
  - Toronto, Ontario
  - Sainte-Foy, Quebec
  - Hamilton Ontario
- Chile (3):
  - Rancagua
  - Santiago
  - Temuco IX
- Germany (6):
  - Berlin
  - Cologne
  - Hamburg
  - Hanover
  - Leipzig
  - Rostock
- Budepest, Hungary
- Monterrey, Mexico
- New Zealand (3):
  - Auckland
  - Rotorua
  - Timaru
- Poland (4):
  - Elblag
  - Kalisz
  - Szczecin
  - Warsaw
- South Korea (4):
  - Anyang
  - Daegu
  - Pusan
  - Seoul
- Kaohsiung County, Taiwan

REFERENCES:
- [Derived] Leu JH, Adedokun OJ, Gargano C, Hsia EC, Xu Z, Shankar G. Immunogenicity of golimumab and its clinical relevance in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. Rheumatology (Oxford). 2019 Mar 1;58(3):441-446. doi: 10.1093/rheumatology/key309. PMID 30412238
- [Derived] George MD, Ostergaard M, Conaghan PG, Emery P, Baker DG, Baker JF. Obesity and rates of clinical remission and low MRI inflammation in rheumatoid arthritis. Ann Rheum Dis. 2017 Oct;76(10):1743-1746. doi: 10.1136/annrheumdis-2017-211569. Epub 2017 Jun 12. PMID 28606966
- [Derived] Kay J, Fleischmann R, Keystone E, Hsia EC, Hsu B, Zhou Y, Goldstein N, Braun J. Five-year Safety Data from 5 Clinical Trials of Subcutaneous Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis. J Rheumatol. 2016 Dec;43(12):2120-2130. doi: 10.3899/jrheum.160420. Epub 2016 Nov 1. PMID 27803138
- [Derived] Mack ME, Hsia E, Aletaha D. Comparative Assessment of the Different American College of Rheumatology/European League Against Rheumatism Remission Definitions for Rheumatoid Arthritis for Their Use as Clinical Trial End Points. Arthritis Rheumatol. 2017 Mar;69(3):518-528. doi: 10.1002/art.39945. PMID 27696724
- [Derived] Baker JF, Conaghan PG, Smolen JS, Aletaha D, Shults J, Emery P, Baker DG, Ostergaard M. Development and validation of modified disease activity scores in rheumatoid arthritis: superior correlation with magnetic resonance imaging-detected synovitis and radiographic progression. Arthritis Rheumatol. 2014 Apr;66(4):794-802. doi: 10.1002/art.38304. PMID 24757132
- [Derived] Keystone EC, Genovese MC, Hall S, Miranda PC, Bae SC, Palmer W, Wu Z, Xu S, Hsia EC. Golimumab in patients with active rheumatoid arthritis despite methotrexate therapy: results through 2 years of the GO-FORWARD study extension. J Rheumatol. 2013 Jul;40(7):1097-103. doi: 10.3899/jrheum.120584. Epub 2013 May 15. PMID 23678153
- [Derived] Genovese MC, Han C, Keystone EC, Hsia EC, Buchanan J, Gathany T, Murphy FT, Wu Z, Parasuraman S, Rahman MU. Effect of golimumab on patient-reported outcomes in rheumatoid arthritis: results from the GO-FORWARD study. J Rheumatol. 2012 Jun;39(6):1185-91. doi: 10.3899/jrheum.111195. Epub 2012 Apr 15. PMID 22505702
- [Derived] Visvanathan S, Rahman MU, Keystone E, Genovese M, Klareskog L, Hsia E, Mack M, Buchanan J, Elashoff M, Wagner C. Association of serum markers with improvement in clinical response measures after treatment with golimumab in patients with active rheumatoid arthritis despite receiving methotrexate: results from the GO-FORWARD study. Arthritis Res Ther. 2010;12(6):R211. doi: 10.1186/ar3188. Epub 2010 Nov 17. PMID 21083889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 444 participants were enrolled at 60 sites in 12 countries.
Groups:
- Group 1: Placebo + Methotrexate: Placebo subcutaneous (SC) injections every 4 weeks from Week 0 to Week 20 (early escape at Week 16); Methotrexate - 15 to 25mg weekly from Week 0 up to 5 yrs; Golimumab - if early escape, 50mg SC injections every 4 weeks from Week 16 up to 5 years; Golimumab - 50 mg SC injections every 4 weeks from Week 24 up to 5 yrs (unless early escape); Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100mg and from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 2: Golimumab 100 mg + Placebo: Golimumab 100 mg SC injections every 4 weeks from Week 0 up to 5 yrs; Placebo - 7 to 10 capsules weekly during blinded period (or Week 16 if early escape); Methotrexate - if early escape, 15 to 25mg weekly from Week 16 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 3: Golimumab 50 mg + Methotrexate: Golimumab 50 mg SC injections every 4 weeks from Week 0 up to 5 yrs (unless early escape at Week 16); Methotrexate - 15 to 25 mg weekly from Week 0 up to 5 years; Golimumab - if early escape, 100 mg SC injections every 4 weeks from Week 16 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to100mg and from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 4: Golimumab 100 mg + Methotrexate: Golimumab100 mg SC injections every 4 weeks from Week 0 up to 5 yrs; Methotrexate - 15 to 25 mg weekly from Week 0 up to 5 yrs; Methotrexate - Dr's discretion, weekly dose adjusted after unblinding; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
Period: Overall Study
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate
Started | 133 | 133 | 89 | 89
Completed | 90 | 92 | 72 | 59
Not Completed | 43 | 41 | 17 | 30
Not completed — Death | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 1 | 1
Not completed — Adverse Event | 23 | 18 | 9 | 14
Not completed — Unsatisfactory therapeutic effect | 4 | 11 | 4 | 6
Not completed — Discontinued oral study agent | 0 | 1 | 0 | 0
Not completed — Other | 13 | 7 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Total
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.96) | 50 (11.47) | 50.3 (10.98) | 50 (10.78) | 50.4 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 105 | 72 | 72 | 358
  Male | 24 | 28 | 17 | 17 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved American College of Rheumatology (ACR) 20 Response at Week 14
Description: ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain of pain by the Visual Analogue Scale (VAS) (0-10 cm) b.Patient's Global Assessment of Disease activity VAS (0-10 cm) c. Physician's Global Assessment of Disease Activity VAS (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein.
Time Frame: Week 14
Population: All participants randomly assigned to each treatment group
Measure: Number; unit: Participants
Groups:
- Combined Golimumab + Methotrexate: Combines Group 3 (golimumab 50 mg + methotrexate) and Group 4 (golimumab 100 mg + methotrexate)
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Participants | 44 | 59 | 49 | 50 | 99
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups I vs III and Groups I vs IV at 0.05 level of significance. Assuming greater than 90 % power, ACR 20 response for Group I, Group III and Group IV (120, 80, and 80 participants, respectively) as 35 % for Group I and 55 % for Groups III and IV; Test type: Superiority or Other; p < 0.001, Chi-squared — The positive test is defined if the comparison between combined golimumab+MTX and Group 1 is significant at the 0.05, and at least one of the pair-wise comparisons is also significant at the 0.05
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups I vs III and Groups I vs IV at 0.05 level of significance. Samples of sizes 120, 80, 80 patients in Group I, III, and IV provide >90% power assuming 35% response in Group I and 55% ACR 20 response in golimumab groups(III & IV); Test type: Superiority or Other; p = 0.001, Chi-squared
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Null hypothesis: No difference between Group II and Group I with respect of ACR 20 at Wk 14. Superiority of golimumab alone vs MTX alone will be demonstrated if 2-sided test is significant. Sample of 120 patients in each Group I & II provides >85% power assuming 35% ACR 20 response in Group I and 55% ACR 20 in Group II; Test type: Superiority or Other; p = 0.059, Chi-squared — This null hypothesis is tested only if a positive test for null hypothesis Statistical Analysis 1

2. Secondary Outcome: Number of Participants With Disease Activity Index Score 28 (DAS 28) Using C-reactive Protein (CRP) Response at Week 14
Description: DAS 28 using CRP is an index to measure the disease activity in participants with rheumatoid arthritis which combines tender joint count (28 joints), swollen joint count (28 joints), CRP value, and participant's global assessment of disease activity (using a Visual Analog Scale of 0 to 100 mm). The DAS 28 score ranges from 0 (best) to 10 (worst). Participants are considered to have a DAS 28 response if they have a score of <= 3.2 (good response) or > 3.2 to 5.1 (moderate response).
Time Frame: Week 14
Population: All participants randomly assigned to each treatment group
Measure: Number; unit: Participants
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Participants | 67 | 84 | 64 | 67 | 131
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p = 0.001, Chi-squared
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.035, Chi-squared

3. Primary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Week 24
Description: HAQ is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). The average score across the functional areas yields an overall HAQ score which ranges from 0 (no disability) to 3 (completely disabled).
Time Frame: Baseline (Week 0) and Week 24
Population: All participants randomly assigned to each treatment group
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Units on a scale | 0.1250 [-0.1250 to 0.3750] | 0.1250 [-0.2500 to 0.6250] | 0.3750 [0.1250 to 0.7500] | 0.5000 [0.1250 to 0.7500] | 0.4375 [0.1250 to 0.7500]
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Null hypothesis: No difference in HAQ response at Wk 24 comparing Groups I and Combined Golimumab + Methotrexate (MTX) at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores. — The positive test is defined if the comparison between combined golimumab+MTX and Group I is significant at the 0.05, and at least one of the pair-wise comparisons is also significant at the 0.05
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Null hypothesis: No difference in HAQ response at Wk 24 comparing Groups I and III at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Null hypothesis: No difference in HAQ response at Wk 24 comparing Groups I and IV at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Null hypothesis: No difference in HAQ response at Wk 24 comparing Groups I and II at 0.05 level of significance; Test type: Superiority or Other; p = 0.240, ANOVA on van der Waerden normal scores

4. Secondary Outcome: Number of Participants Who Achieved American College of Rheumatology 20 (ACR 20) Response at Week 24
Description: An ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain (VAS) (0-10 cm) b.Patient's Global Assessment of Disease activity (VAS) (0-10 cm) c. Physician's Global Assessment of Disease Activity (VAS) (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein (CRP).
Time Frame: Week 24
Population: All participants randomly assigned to each treatment group
Measure: Number; unit: Participants
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Participants | 37 | 47 | 53 | 53 | 106
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.187, Chi-squared

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Week 14
Description: The HAQ is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). The average score across the functional areas yields an overall HAQ score which ranges from 0 (no disability) to 3 (completely disabled).
Time Frame: Baseline (Week 0) and Week 14
Population: All participants randomly assigned to each treatment group
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Units on a scale | 0.1250 [-0.1250 to 0.3750] | 0.2500 [-0.1250 to 0.6250] | 0.3750 [0.1250 to 0.7500] | 0.3750 [0.1250 to 0.6250] | 0.3750 [0.1250 to 0.7500]
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden noramal
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.097, ANOVA on van der Waerden normal scores

6. Secondary Outcome: Change From Baseline in Total Van Der Heijde Modified Sharp (vdH-S) Score at Week 24
Description: The vdH-S score is the sum of joint erosion score and joint-space narrowing (JSN) score. The total score ranges from 0 (best) to 448 (worst) with higher scores indicating more joint damage.
Time Frame: Baseline (Week 0) and Week 24
Population: All participants randomly assigned to each treatment group
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 133 | 133 | 89 | 89 | 178
Units on a scale | 0.00 (2.354) [0.00 to 0.50] | 0.00 (1.598) [0.00 to 0.50] | 0.00 (2.740) [0.00 to 0.50] | 0.00 (1.342) [0.00 to 0.50] | 0.00 (2.159) [0.00 to 0.50]
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p = 0.551, ANOVA on van der Waerden normal
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p = 0.953, ANOVA on van der Waerden normal scores
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p = 0.293, ANOVA on van der waerden normal scores
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.361, ANOVA on van der Waerden normal scores

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 years
Description: All patients randomized to the "Placebo + Methorexate" arm at baseline received golimumab at Week 16 (early escape) or Week 24 (cross over). 5-year safety data are presented according to the dose of golimumab received during the study. 10 patients did not receive any treatment with golimumab and are not included in the 5-year safety data.
Groups:
- Group 1: Golimumab 50 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 50 mg injections only during the study. Participants also received methotrexate capsules throughout the study.
- Group 2: Golimumab 100 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 100 mg injections only during the study. Participants also received either methotrexate or placebo capsules throughout the study.
- Group 3: Golimumab 50 and 100 mg SC Injections: Participants who were treated with golimumab and received at least one injection of both golimumab 50 mg and golimumab 100 mg during the study. Participants also received either methotrexate or placebo capsules throughout the study.
Arm/Group | Group 1: Golimumab 50 mg SC Injections Only | Group 2: Golimumab 100 mg SC Injections Only | Group 3: Golimumab 50 and 100 mg SC Injections
Serious Adverse Events (participants affected / at risk) | 33/105 | 84/184 | 55/145
Other Adverse Events (participants affected / at risk) | 96/105 | 160/184 | 118/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg SC Injections Only (N=105) | Group 2: Golimumab 100 mg SC Injections Only (N=184) | Group 3: Golimumab 50 and 100 mg SC Injections (N=145)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 1 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Dressler's Syndrome (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 2 | 0 | 2
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 1 | 0
Scotoma (Eye disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0
Parotid Gland Enlargement (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 1
Necrosis (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 5 | 3
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Anti-Neutrophil Cytoplasmic Antibody Positive Vasculitis (Immune system disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 0 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 2 | 0
Arthritis Infective (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 4 | 1
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 1 | 0
Disseminated Tuberculosis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Empyema (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Incision Site Cellulitis (Infections and infestations) | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 1 | 0
Peritoneal Tuberculosis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3 | 2
Pneumonia Primary Atypical (Infections and infestations) | 0 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 5 | 1
Septic Arthritis Staphylococcal (Infections and infestations) | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Tuberculous Pleurisy (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0
Vulval Cellulitis (Infections and infestations) | 0 | 0 | 1
Abdominal Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Brain Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Column Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Weight Decreased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint Destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 1
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Axonal Neuropathy (Nervous system disorders) | 0 | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Paresis (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Breast Calcifications (Reproductive system and breast disorders) | 1 | 0 | 0
Breast Enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Menopausal Symptoms (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic Adhesions (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal Cord Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0
Hypertensive Emergency (Vascular disorders) | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg SC Injections Only (N=105) | Group 2: Golimumab 100 mg SC Injections Only (N=184) | Group 3: Golimumab 50 and 100 mg SC Injections (N=145)
Anaemia (Blood and lymphatic system disorders) | 5 | 11 | 7
Abdominal Pain (Gastrointestinal disorders) | 3 | 11 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 13 | 15
Diarrhoea (Gastrointestinal disorders) | 16 | 24 | 11
Dyspepsia (Gastrointestinal disorders) | 7 | 11 | 4
Gastritis (Gastrointestinal disorders) | 7 | 9 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 6 | 8
Nausea (Gastrointestinal disorders) | 9 | 23 | 11
Fatigue (General disorders) | 11 | 9 | 3
Injection Site Erythema (General disorders) | 4 | 20 | 3
Oedema Peripheral (General disorders) | 2 | 10 | 9
Bronchitis (Infections and infestations) | 18 | 27 | 28
Fungal Skin Infection (Infections and infestations) | 6 | 2 | 2
Gastroenteritis (Infections and infestations) | 4 | 11 | 7
Herpes Zoster (Infections and infestations) | 9 | 11 | 10
Influenza (Infections and infestations) | 4 | 11 | 9
Nasopharyngitis (Infections and infestations) | 15 | 35 | 24
Oral Herpes (Infections and infestations) | 4 | 9 | 11
Pharyngitis (Infections and infestations) | 13 | 20 | 25
Rhinitis (Infections and infestations) | 7 | 5 | 3
Sinusitis (Infections and infestations) | 6 | 20 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 39 | 64 | 39
Urinary Tract Infection (Infections and infestations) | 9 | 20 | 20
Contusion (Injury, poisoning and procedural complications) | 5 | 13 | 8
Alanine Aminotransferase Increased (Investigations) | 8 | 19 | 11
Aspartate Aminotransferase Increased (Investigations) | 5 | 17 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 14 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 18 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 22 | 20
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 10 | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 10 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 10 | 6
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 13 | 22 | 15
Headache (Nervous system disorders) | 13 | 22 | 20
Depression (Psychiatric disorders) | 1 | 10 | 10
Insomnia (Psychiatric disorders) | 3 | 11 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 35 | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 19 | 15
Skin Lesion (Skin and subcutaneous tissue disorders) | 8 | 6 | 2
Hypertension (Vascular disorders) | 8 | 25 | 21

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days